CLINICAL TRIAL: NCT06264583
Title: Euro-HDV:Epidemiology and Clinical Course in Patients With HIV and Hepatitis B/D -Coinfection
Brief Title: HDV-Europe: Prevalence and Outcome of HDV in HIV/HBV Coinfection
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Collaborators: Swiss HIV Cohort Study (Network); ICONA Cohort (Unknown); Amsterdam UMC (Other); Royal Free Hospital NHS Foundation Trust (Other); King's College London (Other); University Hospital of Cologne (Other); Goethe University (Other); Heinrich-Heine University, Duesseldorf (Other); University Hospital, Essen (Other); ICH Hamburg (Unknown); Praxiszentrum Hohenstaufenring Köln (Unknown); Sorbonne University (Other); Henri Mondor University Hospital (Other); Hospital Universitario Infanta Leonor (Other); Hospital General Universitario Gregorio Marañon (Other); GEPCOI (Portuguese Group of Coinfection) (Unknown)
Responsible Party: Principal Investigator, Jürgen Rockstroh, MD, PhD, Head of Infectious Diseases, University Hospital, Bonn
Other Study IDs: IN-DE-980-6998
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hepatitis D
Keywords: HIV; hepatitis B; hepatitis delta; liver disease associated death
MeSH Terms: conditions — Hepatitis D; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: HDV screening — 1. Analyze the rate of HDV-testing and evaluate the prevalence of HDV-infection by testing.

SUMMARY:
The aim of this project is to set up a cross-sectional cohort study (France, Germany, The Netherlands, Poland, Spain, Switzerland, Italy, United Kingdom and Portugal) to assess the implementation of EACS guidelines for HDV-testing among PLWH with positive HbsAg and thereby evaluate the prevalence of HDV infection among HIV/HBV-coinfected in 2023, as well as corresponding risk factors. In addition to the testing itself, this study will also set up a cohort and databasee for future HDV studies among PLWH, including clinical, virological und laboratory parameters.

1. Analyze the rate of HDV-testing and evaluate the prevalence of HDV-infection by testing.

   1. Evaluation of former screening of HDV by assessing existing data at study sites.
   2. Determination of the HDV prevalence in European PLWH and HBV coinfection.
2. Setting up a database of all PLWH with HBV/HDV coinfection

   1. Analysis of transmission risk factors for HDV coinfection
   2. Asses the rate of HDV positive patients with ongoing HDV replication.
   3. Define the liver disease state by APRI score, fibroscan, ultrasound and routine laboratory test results.

DETAILED DESCRIPTION:
Background Hepatitis D is caused by a defective RNA-virus, that is known to be among the smallest human pathogenic viruses. As it partly shares the viral entry into hepatocytes with HBV, a coinfection is mandatory (1). Besides a simultaneous infection with HBV and HDV, it might also occur in the sense of a superinfection to a preexisting HBV-infection (2). Though most of the acute infections recover spontaneously, a progression to chronic disease is well described (3). The persistence of HDV leads to an accelerated fibrosis progression and eventually to cirrhosis and an increased risk of developing hepatocellular carcinoma (HCC) as well (4, 5). With the widely established feasibility of immunization against viral Hepatitis B, numbers of HDV-infection in high-income countries are quite low. Nevertheless, the burden of chronic HDV-infection worldwide is high, as different studies estimate the number of patients from 12 million to up to 72 million (6-8).

In the subgroup of people living with HIV (PLWH), who are at increased risk for acquiring viral hepatitis in general, rates of HDV infection have been reported between 10%-20% of HIV/HBV-coinfected people, with variations according to region as well as transmission group. Particularly, early in the HV epidemic higher rates of HDV have been reported for HIV/HBV coinfected drug users. More recently, a shift from people who acquired HIV through drug injection (PWID) to men who have sex with men (MSM) has been reported with HDV coinfection rates of around 8% (9). Common for all PLWH with HBV/HDV-coinfection is a more rapid progression in liver disease (10), resulting in increased rates of decompensated cirrhosis and higher mortality (11, 12). Therefore, mandatory screening for HDV was implemented into current EACS guideline recommendations. However, there is still a lack of testing in daily routine, even at sites where testing is easily accessible and reimbursed. Moreover, most PLWH who are coinfected with HBV are tested at initial HBV diagnosis, but after being put on antiretroviral treatment, which usually includes a tenofovir-based therapy a follow-up testing of HDV does not take place routinely.

Objective The aim of this project is to set up a cross-sectional cohort study (France, Germany, The Netherlands, Poland, Spain, Switzerland, Italy, United Kingdom and Portugal) to assess the implementation of EACS guidelines for HDV-testing among PLWH with positive HbsAg and thereby evaluate the prevalence of HDV infection among HIV/HBV-coinfected in 2023, as well as corresponding risk factors. In addition to the testing itself, this study will also set up a cohort and databasee for future HDV studies among PLWH, including clinical, virological und laboratory parameters.

1. Analyze the rate of HDV-testing and evaluate the prevalence of HDV-infection by testing.

   1. Evaluation of former screening of HDV by assessing existing data at study sites.
   2. Determination of the HDV prevalence in European PLWH and HBV coinfection.
2. Setting up a database of all PLWH with HBV/HDV coinfection

   1. Analysis of transmission risk factors for HDV coinfection
   2. Asses the rate of HDV positive patients with ongoing HDV replication.
   3. Define the liver disease state by APRI score, fibroscan, ultrasound and routine laboratory test results.

Cohort Design and Methods General In this multi-center cohort study patients with documented HIV/HBV-coinfection (2 measurements of positive HBsAg > 6month interval and Anti-HBc-positive) will be evaluated for past HDV screening (last 24 months).

Eligible participants must be 18 years of age or older.

Methods:

* HDV-replication will be measured by commercially used PCR-testing kits. The proportion of HDV serological positive individuals with ongoing viral replication will be determined. This will be collected for all patients with positive HDV serology.
* The liver disease stage, which is expressed by the fibrosis stage, will be determined by APRI score. Furthermore, other non-invasive imaging techniques, including standard ultrasound as well as Fibroscan will be used where available to evaluate the degree of liver disease. In addition, standard laboratory parameters (see, eCRF codebook, annex xyz), which are part of the routine testing among PLWH control visits, will be documented. Changes over time will be evaluated and put in relation to medical imaging, as far as available.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-infection confirmed by HIV-ELISA
* Chronic HBV Infection confirmed by d HBV HBsAg-testing (2 measurements of positive HBsAg > 6month interval).

Exclusion Criteria:

* PLWH with a cleared HBV-infection (anti-HBc or anti-HBc and anti-HBs antibody positive will be considered as HIV-monoinfected persons.
* Individuals younger than 18 years of age
* Patients with any social condition or living circumstances which may interfere with the conduct of the study, as anticipated by the investigator, such as incapacity to adequately understand the study content or not willing to cooperate will be excluded from the study. -For France, patients without adequate social security will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To secure representative data, each cohort or clinic network will aim to enroll a sample size of at least 20% of all HIV/HBV-coinfected individuals in each country. The overall number of participants is planned to reach at least 8000 HIV/HBV-coinfected persons. With an estimated 800.000 PLWH in the following 9 countries: Spain 150.00, France 190.000, Germany 93.000, England 106.000, Portugal 61.000, Italy 140.000, Poland 20.000, Switzerland 16.000, Netherlands 24.000, and an estimated HBV-Prevalence of 5%, this would lead to a cohort of around 40.000 HIV/HBV coinfected individuals. According to current data, 20% of HIV/HBV-coinfected PLWH are expected to have an HDV-infection, which should add up to 8000 individuals that would be needed to be studied.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
HDV prevalence in HIV/HBV coinfection | all data collected in 2023
  percentage of HDV seropositive individuls with HIV/HBV coinfection

SECONDARY OUTCOMES:
Degree of liver disease in pateints with HIV/HBV/HDV triple infection | all data collected in 2023
  assess liver fibrosis stage

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Rockstroh, MD, Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Collected data will be analyzed, evaluated and presented in an anonymous form, ensuring confidentiality of patient data towards third parties.

REFERENCES:
- [Background] Botelho-Souza LF, Vasconcelos MPA, Dos Santos AO, Salcedo JMV, Vieira DS. Hepatitis delta: virological and clinical aspects. Virol J. 2017 Sep 13;14(1):177. doi: 10.1186/s12985-017-0845-y. PMID 28903779

DOCUMENTS (1):
  • Study Protocol (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT06264583/Prot_000.pdf